CLINICAL TRIAL: NCT04552262
Title: A Randomized, 2-way Crossover, Placebo-controlled, Double-blind Study to Evaluate Effects of Single Oral Doses of BAY 2327949 on Renal Perfusion in Participants With Moderate Chronic Kidney Disease
Brief Title: Study to Learn More About the Effect of a New Drug Called BAY2327949 on the Blood Flow Through Kidneys in Adult Participants With Moderate Chronic Kidney Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19748; 2019-003569-17 (EudraCT Number)
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Moderate Chronic Kidney Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY2327949 / Placebo (Experimental): Each participant will receive two treatments: a single dose of 90 mg BAY 2327949 (Treatment A) and a single dose of placebo to BAY 2327949 (Treatment B), with a washout period of at least 7 days before the second treatment.
  Interventions: Drug: BAY2327949
- Placebo / BAY2327949 (Experimental): Each participant will receive two treatments: a single dose of 90 mg BAY 2327949 (Treatment A) and a single dose of placebo to BAY 2327949 (Treatment B), with a washout period of at least 7 days before the second treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY2327949 — Single dose of 90 mg BAY2327949
  Arms: BAY2327949 / Placebo
Drug: Placebo — Single dose of placebo to BAY 2327949
  Arms: Placebo / BAY2327949

SUMMARY:
Researchers in this study want to learn more about the effect of a new drug called BAY2327949 on the blood flow through kidneys in adult participants with moderate long lasting kidney disease. It is thought that, in long lasting kidney disease, blood flow through the kidney tissue is changed, and that some parts of the kidney may receive less oxygen and nutrients because of this. BAY2327949 is a new drug under development with a goal to modify how much blood is flowing through kidneys. It works by binding to and blocking proteins that can regulate blood flow through the kidneys.

Participants in this study will receive 3 tablets of BAY2327949 once and 3 tablets of Placebo once (a placebo looks like a drug but does not have any medicine in it). Both BAY2327949 and Placebo will be taken orally. And after taking each of them, participants will undergo a Magnetic Resonance Imaging (MRI) scanning for 60 to 90 minutes to assess the blood flow to kidneys. MRI is an examination of parts of the body (in this case the kidney) which provides images of these regions. Blood samples will be collected from the participants to check the general health and look at how the study drug is working in the body and how the body affects the study drug. Participants will visit the hospital or clinic about 4 times in total, and the observation for each participant will not more than 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 75 years of age inclusive, at the time of signing the informed consent
* Clinical diagnosis of CKD for at least 6 months, with eGFR ≥30 mL/min/1.73 m2 but <60 mL/min/1.73 m2 (eGFR will be estimated at study site from serum creatinine using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
* Copeptin level of ≥10 pmol/L at the screening visit
* Men or confirmed postmenopausal women (documented by medical report verification and defined as exhibiting spontaneous amenorrhea for at least 12 months before screening or as exhibiting spontaneous amenorrhea for 6 months before screening with documented serum follicle-stimulating hormone [FSH] levels >40 mIU/mL) or women without childbearing potential based on surgical treatment 6 weeks before screening such as bilateral tubal ligation, bilateral oophorectomy or hysterectomy (documented by medical report verification).

Sexually active men, who have not been surgically sterilized, must agree to use 2 reliable and acceptable methods of contraception simultaneously (whereby one method has to be applied in the man and one method in the female partner), and not to act as sperm donor. This applies for the time period between signing of the informed consent form (ICF) and 12 weeks after the last administration of study drug.

Acceptable methods of contraception include, but are not limited to, (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception.

* Participants must be able to meet the requirements of the MRI scan (e.g. physically able to fit into the scanner)
* If patient is taking loop diuretics, must be able to discontinue loop diuretics in the morning of Visit 2 and Visit 3.

Exclusion Criteria:

* Known acute kidney diseases (incl. kidney stones) or renal conditions that in the opinion of the investigator are expected to significantly change in intensity over the study period
* Clinical diagnoses of heart failure and persistent symptoms (New York Heart Association class III - IV)
* Systolic blood pressure >160 mmHg, or diastolic blood pressure ≥100 mmHg
* Stroke, transient ischemic cerebral attack, acute coronary syndrome, hospitalization for worsening heart failure or unplanned/emergency hospitalization in the last 3 months prior to randomization
* Renal allograft in place
* Hepatic insufficiency classified as Child-Pugh B or C, or active hepatitis B or C at Visit 1.
* Active malignancy aside from treated squamous cell or basal cell carcinoma of the skin
* Dialysis for acute renal failure within the previous 6 months prior to randomization
* Indication for immunosuppressants, receiving cytotoxic therapy, immunosuppressive therapy, or other immunotherapy within 6 months prior to randomization
* Participant is taking concomitant medication that is:
* - A moderate or strong inhibitor of cytochrome P450 (CYP)3A
* - A moderate or strong inducer of CYP3A
* - A moderate or strong inhibitor of P-glycoprotein transport
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the study intervention
* Previous (i.e. within 3 months prior to randomization) or concomitant participation in another clinical study with the study intervention
* Body mass index (BMI) >35 kg/m²
* Body weight exceeding 120 kg
* Glycosylated hemoglobin (HbA1c) >11% at Visit 1
* History or suggestive of alcohol or substance abuse
* Planned change in dose or schedule of concomitant medication within 4 weeks prior to Visit 1, or planned change during the time course of this study
* Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the participant's safety
* Any other conditions which, in the opinion of the investigator or sponsor, would make the participant unsuitable for inclusion or could interfere with the participant's participation in or completion of the study
* Close affiliation of the participant with the investigational site, e.g. a close relative of the investigator, dependent person (e.g. employee or student of the investigational site)
* Participant is in custody by order of an authority or court of law

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Difference between renal medullary perfusion after administration of BAY 2327949 and placebo as assessed by arterial spin labelling magnetic resonance imaging (ASL-MRI) | Within 2 hours of treatment
  2-way crossover design
  Participants Arm 1:
  Single dose of BAY2327949 + 7 days washout phase + Single dose of Placebo
  Participants Arm 2:
  Single dose of Placebo + 7 days washout phase + Single dose of BAY2327949

SECONDARY OUTCOMES:
Difference between T1 (renal water content) after administration of BAY 2327949 and placebo | Within 2 hours of treatment
  2-way crossover design
  Participants Arm 1:
  Single dose of BAY2327949 + 7 days washout phase + Single dose of Placebo
  Participants Arm 2:
  Single dose of Placebo + 7 days washout phase + Single dose of BAY2327949
  T1 = (renal water content) (unit: ms) acquired during MRI scanning (this parameter will only be obtained at two timepoints, baseline and after the perfusion assessments, and not for all multimodal MRI assessments)
Difference between T2* in the kidney cortex after administration of BAY 2327949 and placebo | Within 2 hours of treatment
  2-way crossover design
  Participants Arm 1:
  Single dose of BAY2327949 + 7 days washout phase + Single dose of Placebo
  Participants Arm 2:
  Single dose of Placebo + 7 days washout phase + Single dose of BAY2327949
  T2 = (unit: ms) acquired during MRI scanning
Difference between T2* in the kidney medulla after administration of BAY 2327949 and placebo | Within 2 hours of treatment
  2-way crossover design
  Participants Arm 1:
  Single dose of BAY2327949 + 7 days washout phase + Single dose of Placebo
  Participants Arm 2:
  Single dose of Placebo + 7 days washout phase + Single dose of BAY2327949
  T2 = (unit: ms) acquired during MRI scanning
Difference between renal cortical perfusion after administration of BAY 2327949 and placebo | Within 2 hours of treatment
  2-way crossover design
  Participants Arm 1:
  Single dose of BAY2327949 + 7 days washout phase + Single dose of Placebo
  Participants Arm 2:
  Single dose of Placebo + 7 days washout phase + Single dose of BAY2327949
Difference between renal arterial flow after administration of BAY 2327949 and placebo | Within 2 hours of treatment
  2-way crossover design
  Participants Arm 1:
  Single dose of BAY2327949 + 7 days washout phase + Single dose of Placebo
  Participants Arm 2:
  Single dose of Placebo + 7 days washout phase + Single dose of BAY2327949
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.